CLINICAL TRIAL: NCT04982354
Title: A Pilot Study of Daunorubicin-cytarabine Liposome (CPX-351) Plus FLT3-inhibitor (Midostaurin) as Induction Therapy for Patients With FLT3 Mutated Acute Myeloid Leukemia Followed by Consolidation With a CD34+-Selected Allograft
Brief Title: Induction Therapy for Patients With FLT3 Mutated Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Could not accrue
Sponsor: Guenther Koehne (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Guenther Koehne, Deputy Director and Chief of Blood and Marrow Transplant, Hematologic Oncology and Benign Hematology, Baptist Health South Florida
Organization: Baptist Health South Florida (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-KOE-003
Record Dates: First submitted 2021-07-13; First posted 2021-07-29 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — CPX-351; midostaurin; Busulfan; Melphalan; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Investigational Treatment (Experimental): Daunorubicin-cytarabine liposome (CPX-351) Plus FLT3-inhibitor (Midostaurin) Induction Therapy followed by Busulfan/Melphalan/Fludarabine Conditioning therapy and CD34+-selected allografts.
  Interventions: Drug: CPX-351; Drug: Midostaurin; Drug: Busulfan; Drug: Melphalan; Drug: Fludarabine; Biological: CD34+ selected allogeneic stem cell transplant from an HLA-compatible donor

INTERVENTIONS:
Drug: CPX-351 — For this trial, patients will be treated with CPX-351 100 (daunorubicin 44 mg/m2 and cytarabine 100 mg/m2) for 3 doses on days 1, 3 and 5 of one and on days 1 + 3 of a second cycle of induction therapy, depending on response obtained following the first induction. Thereafter, up to 2 cycles of consolidation therapy of 2 doses on days 1 and 3 of daunorubicin 29 mg/m2 and cytarabine 65 mg/m2 will be administered to the patients.
Drug: Midostaurin — The FLT3 directed inhibitor, midostaurin, will be given at a dose of 50mg twice daily, starting on day 8 through day 21 of each cycle of CPX-351 until admission for allogeneic stem cell transplant.
  Other Names: Rydapt
Drug: Busulfan — 0.8 mg/kg/dose every six hours x 12 doses administered intravenously
  Other Names: Myleran
Drug: Melphalan — 70 mg/m2/day x 2 doses administered intravenously
  Other Names: Alkeran
Drug: Fludarabine — 25 mg/m2/day x 5 doses administered intravenously
  Other Names: Fludara
Biological: CD34+ selected allogeneic stem cell transplant from an HLA-compatible donor — Allogeneic stem cell transplant infused intravenously

SUMMARY:
This is a pilot study designed to identify the effect of daunorubicin-cytarabine liposome (CPX-351) in combination with a FLT3-inhibitor (midostaurin) as induction and consolidation therapy for patients with high-risk FLT3 mutated acute myeloid leukemia (AML) and subsequent CD34+-selected allogeneic stem cell transplant from HLA compatible related or unrelated donors.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a Karnofsky (adult) Performance Status of at least 70%.
* Patients must have adequate organ function

Exclusion Criteria:

* Female patients who are pregnant or breast-feeding
* Active viral, bacterial or fungal infection
* Patient seropositive for Human Immunodeficiency Virus (HIV-I /II); Human T-Cell Lymphotrophic Virus (HTLV -I /II)
* Presence of leukemia in the Central Nervous System (CNS).

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2031-08-01 (Estimated); Study Completion 2032-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in the complete remission rate | 3, 6, 12 and 24 months
  Assess the complete remission rate following induction therapy with CPX-351 plus midostaurin when administered to patients
Change in Progression Free Survival (PFS) | 3, 6, 12 and 24 months
  to determine the PFS of these patients following allo SCT. To estimate PFS the Kaplan-Meier method will be used.
Change in Overall Survival (OS) | 3, 6, 12 and 24 months
  to determine the OS of these patients following allo SCT. To estimate OS the Kaplan-Meier method will be used.

SECONDARY OUTCOMES:
Change in the rate of Minimal Residual Disease (MRD) negativity | 3, 6, 12 and 24 months
  Ascertain the rate of MRD negativity by next generation sequencing at sequential time post following induction treatment at complete remission prior to allo Stem Cell Transplantation (SCT)
Correlation of Minimal Residual Disease (MRD) | 3, 6, 12 and 24 months
  Correlation of duration of MRD negative status with duration of complete remission of these patients will be assessed using Spearman's correlation with reported p value.

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Koehne, MD. PhD, Principal Investigator — Miami Cancer Institute at Baptist Health of South Florida
Locations (1):
- Miami Cancer Institute at Baptist Health of South Florida, Miami, Florida, United States

REFERENCES:
- See also: Miami Cancer Institute Website — http://baptisthealth.net/cancer-care/home